CLINICAL TRIAL: NCT05915416
Title: The Effect of Child Abuse and Neglect Prevention Program on Awareness Levels and Child Abuse Potential of Pregnant Women: A Randomized Controlled Study
Brief Title: The Effect of Child Abuse and Neglect Prevention Program on Awareness Levels and Child Abuse Potential of Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Damla Özçevik Subaşı, Principal Investigator, Dr, Koç University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KocU-OZCEVIKSUBASI-001
Record Dates: First submitted 2023-06-13; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Child Abuse
Keywords: child abuse; awareness; pregnant; nurse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Researcher and participants could not be blinded due to the nature of the research. Data were coded as 'A' for experiment group and 'B' for control group. Statistical analysis of the coded data was performed by a statistics professional in order to avoid bias in the statistical evaluation of research data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment Group (Experimental): The participants in the experiment group were first administered the pre-test and then CANPP. A Child abuse and neglect Training Booklet was sent to the participants after the pre-test and before the program. Trainings within the scope of CANPP were provided over the Google Meet application in four sessions. A link was sent to the pregnant women via WhatsApp just before the specified training hours so that they could participate in the online training which is carried out individually.
  Interventions: Behavioral: Child Abuse and Neglect Prevention Program
- Control group (No Intervention): Participants in control group does not receive intervention. They were then applied CANPP and were given the training booklet after the finalization the program.

INTERVENTIONS:
Behavioral: Child Abuse and Neglect Prevention Program — The Child Abuse and Neglect Prevention Program was then revised in line with the opinions and suggestions of the experts. Power-point presentations and training booklet prepared for the final form of this program have been prepared in such a way that the content is exactly the same. Training booklet was distributed to the experiment group after the pre-test and to the control group after the re-test. This booklet is designed as a resource that participants can refer to whenever they need it. Trainings were provided online through the Google Meet application, in a total of four sessions with an average of 30 minutes per session. The contents of the trainings are child neglect, physical abuse, emotional abuse and sexual abuse, respectively. Four different power-point presentations, addressing these sub-dimensions, were prepared for training purposes.
  Arms: Experiment Group

SUMMARY:
The aim of this study is to determine the effect of the Child Abuse and Neglect Prevention Program (CANPP) based on Social Cognitive Theory (SCT) on the awareness levels and child abuse potential of pregnant women. This randomized controlled study was conducted between July and December 2022 in a family health center of Aydin/Turkey with the participation a total of 30 pregnant women, who were then distributed into two groups as 15 experiment group and 15 control group pregnant women.The participants in the experiment group were applied SCT-based CANPP whereas no intervention was applied to the control group. Research data were collected before the intervention, one month after the intervention, and three months after the intervention using the Pregnant Data Collection Form, Child Neglect and Abuse Awareness Scale for Parents (CNAASP) and Child Abuse Potential Inventory (CAPI). Chi-Square and Fisher exact tests, independent groups t-test and repeated measures ANOVA test were used in the statistical analysis of the research data.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who agree to participate in the study
* are 18 years of age or older
* who can read and understand Turkish
* who have either a smart phone or a computer
* are between 28+0 and 33+0 weeks of pregnancy

Exclusion Criteria:

* Pregnant women with high risk pregnancy
* who have visual or auditory problems
* who have been diagnosed with mental disorders.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Child Neglect and Abuse Awareness Scale for Parents | one month after the intervention
  Child Neglect and Abuse Awareness Scale for Parents is a 5-point Likert-type scale (1-strongly disagree, 2-disagree, 3-undecided, 4-agree, 5-strongly agree) and consisting of 45 items in total. The scale has 5 sub-dimensions namely General Information (12 items), Physical Abuse (6 items), Emotional Abuse (15 items), Sexual Abuse (8 items), Neglect (4 items). By adding all sub-dimensions, the Child Neglect and Abuse Awareness Scale for Parents total score is calculated. The higher this total score, the higher the awareness of child abuse and neglect.
Child Neglect and Abuse Awareness Scale for Parents | three months after the intervention
  Child Neglect and Abuse Awareness Scale for Parents is a 5-point Likert-type scale (1-strongly disagree, 2-disagree, 3-undecided, 4-agree, 5-strongly agree) and consisting of 45 items in total. The scale has 5 sub-dimensions namely General Information (12 items), Physical Abuse (6 items), Emotional Abuse (15 items), Sexual Abuse (8 items), Neglect (4 items). By adding all sub-dimensions, the Child Neglect and Abuse Awareness Scale for Parents total score is calculated. The higher this total score, the higher the awareness of child abuse and neglect.

SECONDARY OUTCOMES:
Child Abuse Potential Inventory | one month after the intervention
  Child Abuse Potential Inventory used in this study was first developed in 1979 to determine the child abuse potential of adults towards children. Main scale of Child Abuse Potential Inventory is the "abuse scale" (77 items) which measures the child abuse potential of the respondent. Remaining 6 scales (Stress scale, Unhappiness scale, Problems Related to Child and Self scale, Family-Related Problems and Problems Related to Others Scale measure factors related to abuse. Three scales, namely Lie Scale, Random Response Scale and Inconsistency Scale were designed to assess the validity of responses. This study is based on the Child Abuse Potential Inventory 'Abuse Scale'. The cut-off point for abuse scale is 215, but above 166 is considered dangerous. High scores in abuse scale indicate that the respondent has a high potential for child abuse.
Child Abuse Potential Inventory | three month after the intervention
  Child Abuse Potential Inventory used in this study was first developed in 1979 to determine the child abuse potential of adults towards children. Main scale of Child Abuse Potential Inventory is the "abuse scale" (77 items) which measures the child abuse potential of the respondent. Remaining 6 scales (Stress scale, Unhappiness scale, Problems Related to Child and Self scale, Family-Related Problems and Problems Related to Others Scale measure factors related to abuse. Three scales, namely Lie Scale, Random Response Scale and Inconsistency Scale were designed to assess the validity of responses. This study is based on the Child Abuse Potential Inventory 'Abuse Scale'. The cut-off point for abuse scale is 215, but above 166 is considered dangerous. High scores in abuse scale indicate that the respondent has a high potential for child abuse.

CONTACTS AND LOCATIONS:
Locations (1):
- Koç University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No